CLINICAL TRIAL: NCT02149992
Title: Glycemic Impact of Myo-inositol in High Risk and Gestational Diabetic Pregnancies: a Pilot Study
Brief Title: Glycemic Impact of Myo-inositol in Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Duke University (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Amy Valent, DO; Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-1676
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Gestational Diabetes Mellitus as Antepartum Condition
Keywords: gestational diabetes; myoinositol
MeSH Terms: conditions — Diabetes, Gestational | interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myo-inositol, folic acid (Experimental): 1. myo-inositol, oral, 2g, two times per day for 5 total days
  2. folic acid, oral 200 micrograms, two times per day for 7 days
  3. Continuous Glucose Monitoring Surveillance device for 7 days during study period
  4. Capillary glucose monitoring 4 times per day
  Interventions: Dietary Supplement: myo-inositol; Device: Continuous glucose monitoring surveillance; Device: Glucose monitoring

INTERVENTIONS:
Dietary Supplement: myo-inositol — myo-inositol, oral, 2g, twice a day for 5 days total
  Other Names: Inositol
Device: Continuous glucose monitoring surveillance — monitoring device will be placed by experienced research members to the patient on Day 1 and she will continue to wear until Day 7. This device monitors overall glycemia every 5 minutes and records the information, which can be downloaded after discontinued.
  Other Names: Medtronic CGMS
Device: Glucose monitoring — patients will use the glucose meter, test strips, and lancets to determine her capillary glucose levels 4 times per day (fasting, and 1 hour post-prandial levels)
  Other Names: OneTouch glucose meter; test strips; lancets

SUMMARY:
Myo-inositol has been shown to decrease the rate of diabetes in pregnancy in European studies. It is not known exactly how this occurs or what it does to the sugar when the supplement is taken. This study purpose is to look at the patient's sugar levels while taking the supplement to see if the overall levels of sugar go down. We hypothesize that in addition to sugar levels, other hormones influencing diabetes will be altered.

DETAILED DESCRIPTION:
Myo-inositol is important for glucose homeostasis and has been shown to improve insulin sensitivity. This is a prospective cohort pilot study to determine daily glycemic pharmacokinetics and metabolic influences of myo-inositol supplementation using continuous glucose monitoring system (CGMS) and pre- and post-supplement blood work in high risk pregnancies and women diagnosed with gestational diabetes mellitis (GDM). Risk factors include: obesity, previous pregnancy with GDM, family history of diabetes, glucose intolerance, and polycystic ovarian syndrome (PCOS). Women will have a CGMS device placed on day one and begin with 3 days of placebo plus folic acid (400mcg) to determine baseline glycemia and metabolic levels. For the final 4 days, women with take myo-inositol supplementation (4g) plus folic acid (400mcg). The CGMS device will be removed on day 7 when final blood work will be obtained. Self-capillary glucose testing 4 times per day is recorded to calibrate CGMS glucose values. These observations will help determine the effects of myo-inositol on overall mean glucose and other metabolic factors in high risk and GDM patients, identify pharmacokinetic discipline in pregnancy, and develop the groundwork for future prospective clinical trials for the prevention and/or augmentation in treatment GDM.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* singleton
* pregnant females between 20-28 weeks of gestation at time of enrollment PLUS (either of the following)
* High risk including women must have passed routine glucose screening and have greater than or equal to 1 of the following high risk criteria: first degree family member with diabetes mellitus, previous pregnancy with gestational diabetes, PCOS, or body mass index great than or equal to 30.
* Gestational diabetes diagnosed in current pregnancy based on IADPSG or NIH consensus diagnostic recommendation

Exclusion Criteria:

* pre-pregnancy diagnosis of diabetes mellitus
* renal disease
* immunocompromised
* currently taking immunosuppressive medications
* age <13 years old
* non-English speaking
* multifetal gestation.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
overall mean glucose | 7 days
  Difference in overall mean glucose with folic acid alone versus myo-inositol+folic acid supplementation; measured by continuous glucose monitoring system started pre-supplementation and continued for 4 days after supplementation.

SECONDARY OUTCOMES:
metabolic differences | 1,4,7 days
  Metabolic differences (myo-inositol, chiro-inositol, fasting insulin, c-peptide, and adiponectin) pre and post supplementation.

OTHER OUTCOMES:
side effects | day 1,4,7,10
  Through patient surveys, will determine side effect profiles of the supplement
steady state | day 1, 4, 7
  Determine time (days) of supplement required to reach steady state by measuring pre, 1 day post, and at day 4 after supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Valent, DO, Principal Investigator — Test Organization
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States